CLINICAL TRIAL: NCT06813664
Title: A Phase II Open-Label Trial: ctDNA-Guided CURB for OPD mNSCLC on TKI (CURB-TKI)
Brief Title: ctDNA-Guided CURB for OPD mNSCLC on TKI (CURB-TKI)
Acronym: CURB-TKI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-6091
Record Dates: First submitted 2025-01-24; First posted 2025-02-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer; OligoProgressive Metastatic Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decreasing or undetectable ctDNA levels after SBRT/high-dose radiotherapy (Experimental): This group continues the same first-line standard of care or targeted systemic therapy after completion of SBRT.
  Interventions: Radiation: Radiotherapy
- Persistent or increasing ctDNA levels after SBRT/high-dose radiotherapy (Experimental): This group of patients will be switched to a different targeted therapy (second line) or standard of care systemic therapy after completion of SBRT.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — SBRT/high-dose radiotherapy Standard of care targeted therapy
  Arms: Decreasing or undetectable ctDNA levels after SBRT/high-dose radiotherapy
Radiation: Radiotherapy — SBRT/high-dose radiotherapy Second-line targeted therapy
  Arms: Persistent or increasing ctDNA levels after SBRT/high-dose radiotherapy

SUMMARY:
This is an open-label, prospective single arm Phase II trial that investigates the role of ablative stereotactic body radiation therapy (SBRT) in oncogene driven metastatic non-small cell lung cancer (mNSCLC) patients with oligoprogressive disease (OPD) on targeted therapy (TKI) followed by circulating tumor DNA (ctDNA) analysis for tailoring targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Able to do most daily activities (ECOG 0-2).
3. Able and willing to sign an informed consent form to join the study.
4. Metastatic non-small cell lung cancer (NSCLC) with either an EGFR mutation or ALK rearrangement confirmed by imaging and biopsy.
5. Eligible for second-line therapy or targeted treatment (TKI) if in Group B.
6. Willing to give a blood sample for ctDNA analysis.
7. No limit to how many metastatic sites, but up to 5 progressive lesions that do not require immediate treatment.
8. Prior radiation therapy near progressive lesions is allowed if applicable.
9. Cancer lesions must be treatable with specific radiotherapy methods (like SBRT or ablative therapy).
10. Oligoprogressive disease is evaluated independently for each lesion using specific criteria.
11. Stable brain metastases allowed if asymptomatic and do not require corticosteroids.
12. Prior treatment with radiation for oligoprogressive lesions is allowed as long as they remain asymptomatic and re-treatment is possible.
13. Prior non-stereotactic radiation for palliative purposes is allowed, and if the lesion later progresses but is still asymptomatic and does not require immediate therapy, it can count towards the 5 oligoprogressive lesions.
14. Able and willing to complete quality of life and health utility questionnaires in English, French, or Spanish.
15. Accessible for treatment and follow-up.

Exclusion Criteria:

1. More than 5 extracranial sites of progressive disease.
2. Pregnant.
3. Leptomeningeal disease.
4. Serious health issues that prevent radiotherapy, like ataxia-telangiectasia or scleroderma.
5. Prior radiation therapy near the progressive lesion that would prevent treatment with SBRT due to exceeding limits of healthy tissue tolerance.
6. Any psychological, social, or geographic issues that could make it difficult to comply with the study.
7. Any other condition that the investigator believes makes participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free-survival | 1 year
  Progression-free-survival 1 (PFS1) will be determined from the first day of SBRT to oligoprogressive sites to the day of diagnosis of radiological progression in the subsequent imaging (irrespective of change in systemic therapy in group B, essentially second-line) or death

SECONDARY OUTCOMES:
Subsequent progression-free-survival | 1 year
  Subsequent PFS will be calculated from the date of first radiological progression after SBRT to second radiological progression or change to 3rd line systemic therapy or death or loss to follow-up, whichever comes first.
Acute and Late Toxicities | 1 year
  For SBRT combined with TKI (using CTCAE Version 5.0)
Reported Adverse Events | 1 year
  PRO-CTCAE Questionnaire
Quality of Life Outcome | 1 year
  QLQ-LC1 Questionnaire
Quality of Life Outcome | 1 year
  EORTC-QLQ-C30 Questionnaire
Cost-effectiveness | 1 year
  EQ-5D-5L Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Medicine Program, Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada